CLINICAL TRIAL: NCT02293746
Title: Inspire® Upper Airway Stimulation (UAS) System German Post-Market Study: CE Certificate Number 562872
Brief Title: Inspire® Upper Airway Stimulation (UAS) System German Post-Market Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-002
Record Dates: First submitted 2014-11-12; First posted 2014-11-18 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; OSA; neurostimulation; hypoglossal nerve; tongue; upper airway stimulation; surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Inspire Upper Airway Stimulation System
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inspire® UAS System (Other): This is a single-arm study; all participants will be implanted with the Inspire® Upper Airway Stimulation (UAS) System.
  Interventions: Device: Inspire® Upper Airway Stimulation (UAS) System

INTERVENTIONS:
Device: Inspire® Upper Airway Stimulation (UAS) System — This is a single-arm study; all participants will be implanted with the Inspire® Upper Airway Stimulation (UAS) System is a permanent, implantable therapy device, which consists of three implantable components: an IPG, a stimulation lead, and a sensing lead. In addition, the patient receives a remove to activate the therapy.
  Other Names: Inspire® Therapy

SUMMARY:
The purpose of this study is to obtain additional safety and efficacy data on the use of Inspire® therapy for the treatment of subjects with moderate to severe Obstructive Sleep Apnea.

DETAILED DESCRIPTION:
This is a multi-center, prospective, single-arm study conducted under a common implant and follow-up protocol. Each subject will serve as their own control.

The study will collect pre-operative two-night home sleep testing, medical history and subject quality of life measures. Intra- and post- operative procedure data will be collected. Therapy usage and device adjustment data, as well as a subject satisfaction with therapy survey, will be collected for additional analysis.

Post-implant, procedure- and device-related events, QoL questionnaires, therapy usage and device adjustment data will be collected. Sleep study data will collected during the 2-month visit and, if conducted, a 3-month visit using a single night in-lab titration PSGs At 6 and 12 months post-implant, 2-night home sleep testing will be completed. Safety data will be collected throughout the study. Subjects will be exited from the study following the 12-month visits.

The subject population will consist of otherwise healthy men and women that are at least 21 years old and have: 1) Provided written informed consent to participate, 2) Indicated a willingness to comply with study requirements for the specified follow-up duration, 3) Met all inclusion and exclusion criteria of this protocol.

Up to 60 subjects will be implanted at up to 5 sites in Germany.

ELIGIBILITY:
Inclusion Criteria:

1. Likely suffer moderate-to-severe OSA based on history and physical, or have an established diagnosis of OSA (≥ 15 AHI<65) based on a prior sleep test
2. Willing and capable to have stimulation hardware permanently implanted, and to use the patient programmer to activate the stimulation
3. Willing and capable to return for all follow-up visits and conduct sleep studies at home, including the evaluation procedures and filling out questionnaires
4. Willing and capable of providing informed consent

Exclusion Criteria:

Contraindications

1. Any anatomical finding that would compromise the performance of upper airway stimulation, such as the presence of complete concentric collapse of the soft palate
2. Have any condition or procedure that has compromised neurological control of the upper airway
3. Unable or do not have the necessary assistance to operate the patient programmer
4. Pregnant or plan to become pregnant
5. Require magnetic resonance imaging (MRI)
6. Have an implantable device that may be susceptible to unintended interaction with the Inspire system.

   Additional exclusions for study purposes only:
7. Body Mass Index (BMI) of > 35
8. Central + mixed apneas > 25% of the total apnea-hypopnea index (AHI)
9. Any chronic medical illness or condition that contraindicates a surgical procedure under general anesthesia, as judged by the clinical study Investigator
10. Has a terminal illness with life expectancy < 12 months
11. Active psychiatric disease (psychotic illness, major depression, or acute anxiety attacks) which prevents subject compliance with the requirements of the investigational study testing
12. Any other reason the investigator deems subject is unfit for participation in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-12-11 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
Number of Reported SAEs / Procedure & Device Related AEs | 12 months post-implant
  Safety of the therapy will be assessed via the description of all reported SAEs and all procedure- or device-related AEs. Adverse events will be summarized by seriousness, severity, relatedness to the device and/or procedure and temporal relationship to the procedure. No formal statistical hypotheses will be tested. Only device- or procedure-related AEs will be collected in this post-market study.

SECONDARY OUTCOMES:
Change from Baseline OSA at 12 Months | 12 months post-implant
  Frequencies and description statistics will be used to describe the data gathered in this study. A statistical comparison of pre-implant baseline and follow-up data may be performed.
  Efficacy endpoints will evaluate changes in subjects' quality of life (QoL) and Obstructive Sleep Apnea (OSA) severity through:
  1. QoL: Epworth Sleepiness Scale: improvement from baseline to 12 months
  2. QoL: Functional Outcomes of Sleepiness Questionnaire: improvement from baseline to 12 months
  3. OSA Severity: Oxygen Desaturation Index: Reduction at 12 months as compared to baseline.
  4. OSA Severity: Apnea Hypopnea Index: Reduction at 12 months as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Heiser, Dr. med., Principal Investigator — Klinikum rechts der Isar der Technischen Universität München; Joachim T. Maurer, OA Dr. med., Principal Investigator — Universitäts-HNO-Klinik Mannheim; Armin Steffen, PD Dr. med., Principal Investigator — Klinik für HNO-Heilkunde/HNO-Schlaflabor
Locations (3):
- Germany (3):
  - Klinik für HNO-Heilkunde/HNO-Schlaflabor, Lübeck
  - Universitäts-HNO-Klinik Mannheim, Mannheim
  - Klinikum rechts der Isar der Technischen Universität München, München

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Hofauer B, Philip P, Wirth M, Knopf A, Heiser C. Effects of upper-airway stimulation on sleep architecture in patients with obstructive sleep apnea. Sleep Breath. 2017 Dec;21(4):901-908. doi: 10.1007/s11325-017-1519-0. Epub 2017 May 31. PMID 28567688
- [Derived] Heiser C, Edenharter G, Bas M, Wirth M, Hofauer B. Palatoglossus coupling in selective upper airway stimulation. Laryngoscope. 2017 Oct;127(10):E378-E383. doi: 10.1002/lary.26487. Epub 2017 Jan 20. PMID 28105667
- See also: Peer-reviewed publication/results (Laryngoscope 2018) — https://pubmed.ncbi.nlm.nih.gov/28561345/